CLINICAL TRIAL: NCT07147231
Title: A Phase 1 and Randomized Phase 2 Trial of Pidnarulex (CX-5461) and Cemiplimab (REGN2810) in Refractory Microsatellite Stable Colorectal Cancer
Brief Title: Testing the Effectiveness of the Anti-cancer Drug Pidnarulex (CX-5461) in Combination With Another Anti-cancer Drug Cemiplimab (REGN2810), in Treating Refractory Microsatellite Stable Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-06058; NCI-2025-06058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10716 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10716 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2025-08-28; First posted 2025-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Refractory Colorectal Adenocarcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Unresectable Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy; CX 5461

STUDY DESIGN:
Intervention Model Description: In phase 1, patients will be treated with pidnarulex (CX-5461) in combination with cemiplimab (REGN2810) to determine the pidnarulex (CX-5461) RP2D. In phase 2 (randomized), patients will be randomized to receive either pidnarulex (CX-5461) alone or in combination with anti-PD-1, to evaluate the primary endpoint of progression-free survival.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (cemiplimab, pidnarulex) (Experimental): Patients receive cemiplimab IV over 30 minutes on days 1 and 15 of each cycle and pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days for up to 26 cycles of cemiplimab and indefinitely for pidnarulex in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection on study and CT, MRI, or PET/CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pidnarulex; Procedure: Positron Emission Tomography
- Phase II arm I (pidnarulex) (Active Comparator): Patients receive pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and CT, MRI, or PET/CT throughout the trial. Additionally, patients undergo blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pidnarulex; Procedure: Positron Emission Tomography
- Phase II arm II (cemiplimab, pidnarulex) (Experimental): Patients receive cemiplimab IV over 30 minutes on days 1 and 15 of each cycle and pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days for up to 26 cycles of cemiplimab and indefinitely for pidnarulex in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and CT, MRI, or PET/CT throughout the trial. Additionally, patients undergo blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pidnarulex; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Phase II arm I (pidnarulex); Phase II arm II (cemiplimab, pidnarulex)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
  Arms: Phase II arm II (cemiplimab, pidnarulex)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Pidnarulex — Given IV
  Other Names: CX-5461; CX5461; Pol I Inhibitor CX5461; RNA Pol I Inhibitor CX5461
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I/II trial studies the side effects and best dose of pidnarulex when given together with cemiplimab and to see how well it works in treating patients with microsatellite stable (MSS) colorectal cancer (CRC) that does not respond to treatment (refractory). Pidnarulex may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pidnarulex with cemiplimab may be safe, tolerable and/or effective in treating patients with refractory MSS CRC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended phase 2 dose of pidnarulex (CX-5461) with anti-programmed cell death protein 1 (PD-1) in phase 1, and to determine safety and tolerability of pidnarulex (CX-5461) alone, and in combination with anti-PD-1 in phases 1 and 2.

II. To determine the progression-free survival (PFS) of pidnarulex (CX-5461) alone and in combination with anti-PD-1 in patients with refractory liver metastatic microsatellite stable (MSS) colorectal cancer (CRC) associated with replication stress in phase 2.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To compare the objective response rate (ORR) and disease control rate (DCR) of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2.

III. To compare the duration of response (DoR) of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2.

IV. To compare the overall survival (OS) of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2.

V. To evaluate plasma pharmacokinetic (PK) profiles of pidnarulex (CX-5461) alone and in combination with anti-PD-1.

VI. To evaluate the plasma PK profile of cemiplimab. VII. To explore gene signature patterns at baseline or following treatment that may suggest, response to pidnarulex (CX-5461) alone or in combination with anti-PD-1, by whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing in tumor tissue and cell-free deoxyribonucleic acid (DNA) in peripheral blood in phase 2.

EXPLORATORY OBJECTIVES:

I. To evaluate the baseline expression of MYC and CCNE1 in tumor tissue and its association with response to treatment, as identified by immunohistochemistry in phase 2.

II. To evaluate the stimulator of interferon genes (STING) pathway activation and immune cell profile in the tumor at baseline and after treatment with pidnarulex (CX-5461) alone or in combination with anti-PD-1, and its association with response to treatment, as identified by immunohistochemistry in phase 2.

III. To evaluate replication stress at baseline and after treatment, and its association with response to treatment, as identified by immunohistochemistry in phase 2.

IV. To explore pidnarulex (CX-5461) target engagement, as identified by 47S pre-ribosomal ribonucleic acid (rRNA) in-situ hybridization in phase 2.

V. To explore DNA alterations in circulating-tumor deoxyribonucleic acid (ctDNA) and their potential correlation with response to treatment in phase 2.

OUTLINE: This is a phase I, dose-escalation study of pidnarulex in combination with cemiplimab followed by a phase II study.

PHASE I:

Patients receive cemiplimab intravenously (IV) over 30 minutes on days 1 and 15 of each cycle and pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days for up to 26 cycles of cemiplimab and indefinitely for pidnarulex in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection on study and computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT throughout the trial.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and CT, MRI, or PET/CT throughout the trial. Additionally, patients undergo blood sample collection on study.

ARM II: Patients receive cemiplimab IV over 30 minutes on days 1 and 15 of each cycle and pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days for up to 26 cycles of cemiplimab and indefinitely for pidnarulex in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and CT, MRI, or PET/CT throughout the trial. Additionally, patients undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed colorectal adenocarcinoma that is unresectable and/or metastatic and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1
* Patients must have proficient mismatch repair and/or microsatellite stable status
* Phase 2 patients must have at least one liver metastasis at study entry (by imaging and/or histology, per investigator assessment); this metastasis does not need to be measurable
* Phase 2 patients must have local/standard of care tumor molecular testing (tumor tissue or circulating tumor DNA) demonstrating MYC amplification or deleterious/likely deleterious FBXW7 mutation, as defined in the report
* Phase 2 patients must have at least one tumor lesion amenable to biopsy
* Patients must undergo a washout period of 28 days for epidermal growth factor receptor (EGFR) inhibitors, including cetuximab and panitumumab
* Patients must have progressed on or have intolerance to (if eligible and not contraindicated per treating investigator) fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab, and epidermal growth factor receptor (EGFR) inhibitor. These are standard of care treatments for this patient population with proven survival benefit, so it would not be appropriate for patients to enroll in this trial without this criterion being met
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of pidnarulex (CX-5461) in combination with cemiplimab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level of up to 3 mg/dl may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN, (5 × ULN for patients with liver involvement)
* Glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for ≥ 1 month after treatment of the brain metastases
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of that pidnarulex (CX-5461) on the developing human fetus are unknown. Based on its mechanism of action, cemiplimab (REGN2810) can cause fetal harm when administered to a pregnant woman. Animal studies have demonstrated that inhibition of the PD-1/PD-L1 pathway can lead to increased risk of immune-mediated rejection of the developing fetus resulting in fetal death. For these reasons, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) 14 days prior to study entry, for the duration of study participation and for at least 4 months after the last dose of cemiplimab (REGN2810) and 6 months after the last dose of pidnarulex (CX-5461). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women should not breastfeed while taking cemiplimab (REGN2810) for at least 4 months after cessation of treatment, and for pidnarulex (CX-5461), for 6 months after cessation of treatment. Women should not donate eggs for14 days prior to the study, for the duration of study participation, and 6 months after completion of pidnarulex (CX-5461) and cemiplimab (REGN2810). Male patients must also agree to not donate sperm for 14 days prior to the study, for the duration of study participation, and 6 months after completion of pidnarulex (CX-5461) and cemiplimab (REGN2810) administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients with active autoimmune diseases, defined as requiring systemic treatment in the past 2 years with use of disease modifying agents, corticosteroids, or immunosuppressive drugs. Replacement therapy (eg; thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Patients with prior treatment with an RNA polymerase inhibitor, G quadruplex stabilizer, or immunotherapy. This includes prior treatment with a PD-1 or PD-L1 inhibitor agent
* Presence of known photosensitivity disorders

  * Patients who do not agree to use sunglasses and sunscreen (≥ sun protective factor (SPF) 50 to ultraviolet B (UVB) and a high degree of protection against ultraviolet A (UVA) if exposed to sunlight during the study and for 4 weeks after the last dose are not eligible. Patients may also not use sun tanning beds during the study, and within 4 weeks after the last dose
* Patients with a history of cicatricial conjunctivitis or active ocular surface disease (as evaluated by ophthalmologist as needed; routine eye exam for all study participants is not needed)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pidnarulex (CX-5461) and cemiplimab
* Patients who use strong CYP3A4 inhibitors or strong CYP3A4 inducers. Pidnarulex (CX-5461) has been shown to be metabolized primarily by the CYP3A4 enzyme. Inhibitors and substrates of these enzymes can increase pidnarulex (CX-5461) plasma concentrations while inducers of these enzymes can decrease pidnarulex (CX-5461) plasma concentrations
* Patients who are taking corticosteroids at a dose greater than 10 mg of prednisone daily or other immunosuppressive or disease-modifying agents, as this may reduce efficacy of an immunotherapy regimen
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant and lactating women are excluded from this study. The exclusion is based on the potential risk of adverse effects of pidnarulex (CX-5461) on fetal development and newborn health. The safety of pidnarulex (CX-5461) has not been established in pregnant or lactating women, and there is a possibility that the drug could cause harm to the developing fetus or be transferred to the infant through breast milk. Additionally, the physiological changes that occur during pregnancy and lactation could alter the pharmacokinetics and pharmacodynamics of pidnarulex (CX-5461), leading to unpredictable drug exposure and efficacy. There is also an increased risk of immune-mediated rejection of the developing fetus with cemiplimab (REGN2810)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of pidnarulex (CX-5461) with anti-programmed cell death protein 1 (anti-PD-1) (Phase 1) | Up to 28 days
  The Bayesian optimal interval design will be employed to identify the RP2D of pidnarulex (CX-5461) in combination with anti-PD-1.
Incidence of adverse events, serious adverse events, and dose limiting toxicities | Up to 30 days after last dose of study drug
  Will evaluate safety and tolerability of pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phases 1-2. Safety and tolerability will be summarized via descriptive statistics, including adverse events, serious adverse events, and dose limiting toxicities.
Progression-free survival (PFS) (Phase II) | From randomization until disease progression (as assessed by Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1) or death from any cause, whichever occurs first, assessed up to 2 years
  Will evaluate PFS of pidnarulex (CX-5461) alone and in combination with anti-PD-1 in patients with refractory liver metastatic microsatellite stable colorectal cancer associated with replication stress in phase 2. PFS will be compared between the 2 treatment groups following the futility boundary on hazard ratio (HR) derived by using a Hwang-Shih-DeCani spending function with gamma = -2.909. The Kaplan-Meier method will be used to estimate median PFS, PFS rates at different time points, and their 95% confidence intervals (CIs), using the Brookmeyer Crowley's method. The HR and the corresponding two-sided 95% CI will be estimated in a stratified Cox regression model. Stratification factors are consistent with those used at randomization. Subgroup analysis will be performed to assess the consistency of treatment effect across subgroups.

SECONDARY OUTCOMES:
Objective response rate (ORR) (Phase 2) | Up to disease progression or subsequent anticancer therapy, or until the last evaluable tumor assessment in the absence of disease progression, assessed up to 2 years
  Will evaluate the ORR of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2. Defined as the proportion (%) of patients with confirmed complete response (CR) or partial response (PR) as assessed according to RECIST v1.1. ORR will be compared to historical control following Simon's two stage design for the within-arm analysis. The cumulative frequency estimated ORR with corresponding 95% CI will be reported.
Disease control rate (DCR) (Phase 2) | Up to disease progression or subsequent anticancer therapy, or until the last evaluable tumor assessment in the absence of disease progression, assessed up to 2 years
  Will evaluate the DCR of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2.Defined as the proportion (%) of patients with confirmed CR, PR or stable dsiease as assessed according to RECIST v1.1. The cumulative frequency estimated DCR with corresponding 95% CI will be reported.
Duration of response (DOR) (Phase 2) | From the first recorded response (confirmed CR or PR) to the first recorded disease progression (according to RECIST v1.1) or death from any cause, whichever occurs first, assessed up to 2 years
  Will evaluate the DOR of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2. Will be evaluated only for patients who achieve CR or PR. DOR will be summarized descriptively using the Kaplan-Meier method.
Overall survival (OS) (Phase 2) | From randomization until death from any cause, assessed up to 2 years
  Will evaluate the OS of patients treated with pidnarulex (CX-5461) alone and in combination with anti-PD-1 in phase 2. OS will be summarized descriptively using the Kaplan-Meier method.
Pharmacokinetic (PK) parameters of pidnarulex (CX-5461) | Cycle (C) 1 day (D) 1, C1D8, C1D9, C1D15, C2D1, C2D15, C3D1, C6D1, C9D1, C12D1
  Will evaluate the PK parameters of pidnarulex (CX-5461) when given alone and in combination with anti-PD-1, including volume of distribution, area under the curve, maximum serum concentration, serum half-life, and accumulation. Will be reported descriptively. Will be analyzed with both non-compartmental and nonlinear mixed effects approaches. Will also be compared between the randomized arms.
PK parameters of cemiplimab (REGN2810) | C1D1, C1D8, C1D9, C1D15, C2D1, C2D15, C3D1, C6D1, C9D1, C12D1
  Will evaluate the PK parameters of cemiplimab (REGN2810), including clearance. Will be reported descriptively. Will be analyzed with both non-compartmental and nonlinear mixed effects approaches.
Gene signature patterns (Phase 2) | At baseline and 30 days after last dose of study drug
  Will evaluate gene signature patterns at baseline or following treatment that may suggest response to pidnarulex (CX-5461) alone or in combination with anti-PD-1, by whole exome sequencing and ribonucleic acid sequencing in tumor tissue and cell-free deoxyribonucleic acid (DNA) in peripheral blood in phase 2.

OTHER OUTCOMES:
Expression of MYC and CCNE1 (Phase 2) | At baseline
  Will evaluate baseline expression of MYC and CCNE1 in tumor tissue and its association with response to treatment, as identified by immunohistochemistry in phase 2. Will be evaluated and correlated with safety and efficacy outcomes.
Stimulator of interferon genes (STING) pathway activation and immune cell profile (Phase 2) | At baseline and 30 days after last dose of study drug
  Will evaluate STING pathway activation and immune cell profile in the tumor at baseline and after treatment with pidnarulex (CX-5461) alone or in combination with anti-PD-1, and its association with response to treatment, as identified by immunohistochemistry in phase 2. Will be correlated with safety and efficacy outcomes.
Replication stress (Phase 2) | At baseline and 30 days after last dose of study drug
  Will evaluate replication stress at baseline and after treatment, and its association with response to treatment, as identified by immunohistochemistry in phase 2. Will be correlated with safety and efficacy outcomes.
Pidnarulex (CX-5461) target engagement (Phase 2) | Up to 30 days after last dose of study drug
  Will evaluate pidnarulex (CX-5461) target engagement, as identified by 47S pre-ribosomal ribonucleic acid in-situ hybridization in phase 2. Will be correlated with safety and efficacy outcomes.
DNA alterations (Phase 2) | Up to 30 days after last dose of study drug
  Will evaluate DNA alterations in circulating-tumor DNA and their potential correlation with response to treatment in phase 2. Will be correlated with safety and efficacy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Wells A Messersmith, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm